CLINICAL TRIAL: NCT02449018
Title: A Randomized, Double Blind, Placebo Controlled Study to Assess the Safety, Tolerability, Pharmacokinetics and Efficacy of Multiple Doses of QBW251 in Patients With COPD
Brief Title: A Safety, Tolerability and Efficacy Study With QBW251 in COPD Patients With QBW251
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CQBW251X2201
Record Dates: First submitted 2015-03-30; First posted 2015-05-20 (Estimated); Results first posted 2018-04-02 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2018-04

CONDITIONS: Chronic Obstructive Pulmonary Disease, COPD
Keywords: COPD,; chronic bronchitis,; inflammation,; airway,; LCI,; pulmonary function test,; lung function,; controlled clinical trial,; randomized,; airflow,; smoker
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Bronchitis, Chronic; Inflammation | interventions — icenticaftor

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- QBW251 (Experimental): QBW251 will be provided to participants during 70 days
  Interventions: Drug: QBW251
- Placebo (Placebo Comparator): Placebo will be provided to participants during 70 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: QBW251 — QBW251 capsule(s) taken orally twice per day
  Arms: QBW251
Drug: Placebo — Matching placebo capsule(s) taken orally twice per day
  Arms: Placebo

SUMMARY:
To evaluate the efficacy, safety and tolerability of multiple doses of QBW251 vs placebo administered orally, on airway function, lung volume, and quality of life in patients with chronic obstructive pulmonary disease (COPD)

ELIGIBILITY:
Inclusion Criteria: Must have a diagnosis of GOLD II-III chronic obstructive pulmonary disease (COPD); Must have clinical diagnosis of chronic bronchitis; Must be either a current smoker (smoked ≤ 1 pack per day on average for the last 3 months with at least a 10 pack year smoking history) OR an ex-smoker with at least a 10 pack year smoking history; Exclusion Criteria: Must not be receiving chronic, daily, systemic steroids; Must not have severe emphysema (determined by HRCT); Must not have had a COPD exacerbation or respiratory tract infection requiring antibiotics or oral steroids or hospitalization within 6 weeks of screening; Must not be pregnant or nursing or a woman of child bearing potential; Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2015-04-30 (Actual); Primary Completion 2016-12-27 (Actual); Study Completion 2017-01-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (16):
- United States (14):
  - Novartis Investigative Site, Birmingham, Alabama
  - Novartis Investigative Site, Fullerton, California
  - Novartis Investigative Site, Waterbury, Connecticut
  - Novartis Investigative Site, Clearwater, Florida
  - Novartis Investigative Site, Port Orange, Florida
  - Novartis Investigative Site, Tampa, Florida
  - Novartis Investigative Site, Normal, Illinois
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, Huntersville, North Carolina
  - Novartis Investigative Site, Shelby, North Carolina
  - Novartis Investigative Site, Medford, Oregon
  - Novartis Investigative Site, Simpsonville, South Carolina
  - Novartis Investigative Site, Spartanburg, South Carolina
  - Novartis Investigative Site, Union, South Carolina
- Poland (2):
  - Novartis Investigative Site, Lodz
  - Novartis Investigative Site, Sobótka

REFERENCES:
- See also: A Plain Language Trial Summary is available on novartisclinicatrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=223

RESULTS

PARTICIPANT FLOW:
Groups:
- QBW251: QBW251(28 day treatment period) and placebo (42 days, run-in and wash-out periods)
- Placebo: Placebo (70 days, run-in, treatment and wash-out periods)
Period: Overall Study
Arm/Group | QBW251 | Placebo
Started | 64 | 28
Completed | 52 | 26
Not Completed | 12 | 2
Not completed — Abnormal laboratory value | 0 | 1
Not completed — Administrative problems | 1 | 0
Not completed — Adverse Event | 5 | 1
Not completed — Protocol deviation | 4 | 0
Not completed — Patient decision | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | QBW251 | Placebo | Total
Number analyzed (Participants) | 64 | 28 | 92
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.6 (6.61) | 64.9 (7.55) | 64.0 (6.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 9 | 40
  Male | 33 | 19 | 52

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Lung Clearance Index (LCI)
Description: Change from baseline to Day 29 in LCI as measured by multiple breath nitrogen washout (MBNW) technique. MBNW is the time taken to wash out nitrogen while breathing 100% oxygen.
Time Frame: Baseline and Day 29
Population: Pharmacodynamics (PD): analysis set included all patients with available PD data and no major protocol deviations with relevant impact on PD data.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | QBW251 | Placebo
Number analyzed (Participants) | 50 | 24
Days | -0.03 (1.28) | -0.16 (1.15)
Statistical Analysis 1: Comparison: QBW251 vs Placebo; Test type: Superiority; p = 0.130, ANCOVA; Mean Difference (Net) = 0.28, 90% CI 2-sided [-0.24 to 0.79], Standard Deviation 0.31

2. Secondary Outcome: Change From Baseline in FEV1 Pre-bronchodilator
Description: Change From Baseline to Day 29 in FEV1 will be measured by spirometer before bronchodilator administration. Forced Expiratory Volume in 1 Second (FEV1) is the amount of air that can be exhaled in 1 second. All spirometry calibrations and evaluations will follow the recommendations of the American Thoracic Society / European Respiratory Society guidelines for acceptability.
Time Frame: Day 29
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | QBW251 | Placebo
Number analyzed (Participants) | 51 | 23
Liters | 0.04 (0.24) | -0.02 (0.23)

3. Secondary Outcome: Change From Baseline in FEV1 Post-bronchodilator
Description: Change From Baseline to Day 29 in FEV1 will be measured by spirometer after bronchodilator administration. Forced Expiratory Volume in 1 Second (FEV1) is the amount of air that can be exhaled in 1 second. All spirometry calibrations and evaluations will follow the recommendations of the American Thoracic Society / European Respiratory Society guidelines for acceptability.
Time Frame: Day 29
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | QBW251 | Placebo
Number analyzed (Participants) | 51 | 24
Liters | 0.05 (0.21) | -0.02 (0.16)

4. Secondary Outcome: Change From Baseline in FVC Pre Bronchodilator
Description: Change From Baseline to Day 29 in FVC will be measured by spirometer before bronchodilator administration. Forced Vital Capacity (FVC) is the maximum amount of air a person can expel from the lungs after a maximum inhalation. All spirometry calibrations and evaluations will follow the recommendations of the American Thoracic Society / European Respiratory Society guidelines for acceptability. Forced vital capacity (FVC) as a measure of lung function, measured before bronchodilator
Time Frame: Day 29
Population: as for outcome 1
Measure: Least Squares Mean (Standard Deviation); unit: Liters
Arm/Group | QBW251 | Placebo
Number analyzed (Participants) | 51 | 23
Liters | 0.07 (0.05) | 0.01 (0.07)

5. Secondary Outcome: Change From Baseline in FVC Post- Bronchodilator
Description: Change From Baseline to Day 29 in FVC will be measured by spirometer after bronchodilator administration. Forced Vital Capacity (FVC) is the maximum amount of air a person can expel from the lungs after a maximum inhalation. All spirometry calibrations and evaluations will follow the recommendations of the American Thoracic Society / European Respiratory Society guidelines for acceptability. Forced vital capacity (FVC) as a measure of lung function, measured after bronchodilator
Time Frame: Day 29
Population: as for outcome 1
Measure: Least Squares Mean (Standard Deviation); unit: Liters
Arm/Group | QBW251 | Placebo
Number analyzed (Participants) | 51 | 24
Liters | 0.03 (0.04) | 0.01 (0.05)

6. Secondary Outcome: Change From Baseline in TLC
Description: Change From Baseline to Day 29 in TLC will be measured by spirometry. Total lung capacity (TLC) is the volume in the lungs at maximal inflation. All spirometry calibrations and evaluations will follow the recommendations of the American Thoracic Society / European Respiratory Society guidelines for acceptability.
Time Frame: Day 29
Population: as for outcome 1
Measure: Least Squares Mean (Standard Deviation); unit: Liters
Arm/Group | QBW251 | Placebo
Number analyzed (Participants) | 50 | 24
Liters | 0.01 (0.07) | -0.07 (0.10)

7. Secondary Outcome: Change From Baseline in RV
Description: Change From Baseline to Day 29 in RV will be measured by spirometry. Residual volume (RV) is the volume of air remaining in the lungs after a maximal exhalation. All spirometry calibrations and evaluations will follow the recommendations of the American Thoracic Society / European Respiratory Society guidelines for acceptability.
Time Frame: Day 29
Population: as for outcome 1
Measure: Least Squares Mean (Standard Deviation); unit: Liters
Arm/Group | QBW251 | Placebo
Number analyzed (Participants) | 48 | 24
Liters | 0.03 (0.07) | -0.02 (0.10)

8. Secondary Outcome: Change From Baseline in FRC
Description: Change From Baseline to Day 29 in FRC will be measured by spirometry. Functional residual capacity (FRC) is the volume in the lungs at the end-expiratory position. All spirometry calibrations and evaluations will follow the recommendations of the American Thoracic Society / European Respiratory Society guidelines for acceptability.
Time Frame: Day 29
Population: as for outcome 1
Measure: Least Squares Mean (Standard Deviation); unit: Liters
Arm/Group | QBW251 | Placebo
Number analyzed (Participants) | 50 | 24
Liters | 0.01 (0.07) | -0.02 (0.09)

9. Secondary Outcome: Change From Baseline in DLCO
Description: Diffusing capacity of the lung for carbon monoxide (DLCO) is the extent to which oxygen passes from the lung to the blood.
Time Frame: Day 29
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: ml/min/mmHg
Arm/Group | QBW251 | Placebo
Number analyzed (Participants) | 42 | 22
ml/min/mmHg | -0.91 (0.24) | -0.25 (0.34)

10. Secondary Outcome: Plasma Concentration of QBW251 by TMax (0-8hours)
Description: Tmax is the time to reach the maximum concentration after drug administration.
Time Frame: Day 1, Day 28
Population: Pharmacokinetics (PK): all patients with at least one available valid PK concentration measurement, who received study drug, and no protocol deviations with relevant impact on PK data. 3 patients had no sufficient concentration data on Day 1 and 2 patients had no concentration data on Days 1 and 28. 7 patients had no concentration data on Day 28
Measure: Median (Full Range); unit: hr
Arm/Group | QBW251
Number analyzed (Participants) | 62
hr
  Day 1: number analyzed (Participants) | 57
  Day 1 | 1.27 [0.983 to 8.03]
  Day 28: number analyzed (Participants) | 53
  Day 28 | 1.98 [0.933 to 7.97]

11. Secondary Outcome: Plasma Concentration of QBW251 by CMax (0-8hours)
Description: Cmax is the observed maximum plasma concentration following drug administration.
Time Frame: Day 1, Day 28
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | QBW251
Number analyzed (Participants) | 62
ng/mL
  Day 1: number analyzed (Participants) | 57
  Day 1 | 1250 (840)
  Day 28: number analyzed (Participants) | 53
  Day 28 | 1640 (916)

12. Secondary Outcome: Plasma Concentration of QBW251 by AUClast (0-8hours)
Description: AUClast is the area under the plasma concentration-time curve from time zero to the time of the last quantifiable concentration.
Time Frame: Day 1, Day 28
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: hr×ng/mL
Arm/Group | QBW251
Number analyzed (Participants) | 62
hr×ng/mL
  Day 1: number analyzed (Participants) | 57
  Day 1 | 3830 (3280)
  Day 28: number analyzed (Participants) | 53
  Day 28 | 6840 (4490)

13. Secondary Outcome: Plasma Concentration of QBW251 by AUC0-12h
Description: AUC 0-12h is the area under the plasma concentration-time curve from time zero to 12 hours.
Time Frame: Day 1, Day 28
Population: PK analysis set: included all patients with at least one available valid PK concentration measurement. Due to practicalities of study conduct PK samples were collected only up to 8 hours. As a result, from noncompartmental analysis AUClast was not calculated up to 12 hours after dosing So this data is not available.
Arm/Group | QBW251 | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events
Groups:
- QBW251 300 mg Bid: QBW251 (28 day treatment period) and placebo (42 days, run-in and wash-out periods)
Arm/Group | Placebo | QBW251 300 mg Bid
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/64
Serious Adverse Events (participants affected / at risk) | 0/28 | 4/64
Other Adverse Events (participants affected / at risk) | 5/28 | 6/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=28) | QBW251 300 mg Bid (N=64)
Vomiting (Gastrointestinal disorders) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=28) | QBW251 300 mg Bid (N=64)
Diarrhoea (Gastrointestinal disorders) | 2 | 2
Nausea (Gastrointestinal disorders) | 2 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety